CLINICAL TRIAL: NCT06206330
Title: The Effect Of Prp (Platelet-Rıch-Plasma) Application On Wound Healing In The Treatment Of Pilonidal Sinus Disease Using Unroofing And Curettage Technique
Brief Title: Effect of Platelet Rich Plasma (PRP) on Healing Time in Patients Following Pilonidal Sinus Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: İsmail Oskay Kaya (Other Government)
Responsible Party: Sponsor-Investigator, İsmail Oskay Kaya, proffesor, Diskapi Yildirim Beyazit Education and Research Hospital
Organization: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 23.08.2021 118/01
Record Dates: First submitted 2023-12-19; First posted 2024-01-16 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Pilonidal Disease; Pilonidal Sinus
Keywords: Platelet rich plasma(PRP); Pilonidal sinus surgery; Healing time
MeSH Terms: conditions — Pilonidal Sinus

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma group (Active Comparator): In this group we applied Platelet rich plasma after the surgery. The surgery was fistulotomy and curettage.
  Interventions: Other: Platelet rich plasma
- Control group (No Intervention): In this group, we did the surgery as fistulotomy and curettage but we did not apply a Platelet rich plasma.

INTERVENTIONS:
Other: Platelet rich plasma — After application of platelet rich plasma after surgery, the patients have examined for infection, hematoma, pain, recurrence and the time of epithelialization of the wound.
  Arms: Platelet rich plasma group

SUMMARY:
Our study was planned as a prospective controlled randomized study. The study was started after the ethics committee approval received from Dışkapı Yıldırım Beyazıt Training and Research Hospital. (23.08.2021 118/01). Two groups of patients were planned in parallel. In the treatment of pilonidal sinus disease, in patients operated on with the fistulotomy and curettage technique, one group was followed up with classical dressing, while the other group was followed up with PRP (platelet-rich-plasma) and classical dressing. Wound infection, hematoma, length of hospital stay, recurrence, pain in the first postoperative week, and time to complete epithelialization of the wound (in days) were evaluated between the two groups.

DETAILED DESCRIPTION:
Our study was planned as a prospective controlled randomized study. The study was started after the ethics committee approval received from Dışkapı Yıldırım Beyazıt Training and Research Hospital. (23.08.2021 118/01). Two groups of patients were planned in parallel. In the treatment of pilonidal sinus disease, in patients operated on with the fistulotomy and curettage technique, one group was followed up with classical dressing, while the other group was followed up with PRP (platelet-rich-plasma) and classical dressing. Wound infection, hematoma, length of hospital stay, recurrence, pain in the first postoperative week, and time to complete epithelialization of the wound (in days) were evaluated between the two groups.

A total of 140 patients, male and female, diagnosed with pilonidal sinus disease in our hospital between November 2021 and November 2022 were included in the study. Patients with acute pilonidal sinus abscess were excluded from the study, but chronic PS(pilonidal sinus) patients who had previously undergone abscess drainage were included in the study.

Patients under 18 years of age, relapsed patients, anemic patients (Hg < 10 mg/dl), thrombocytopenic patients (Plt˂10⁶/ml), patients with a history of radiotherapy-chemotherapy, patients with diabetes and patients using steroids were excluded from the study.

Randomization was performed using the PASS computer program, and according to this randomization, fistulotomy and curettage technique (n=70) was applied to one group and fistulotomy and curettage + PRP (n=70) was applied to the other group.

Demographic information, family history, smoking, presence of abscess drainage, post-drainage antibiotic use, comorbidities, BMI, symptom duration, phenol application, laser epilation, number of sinus pits, presence of secondary orifice, basal PLT(platelet) count, size of the defect after sinus excision, wound infection, hematoma, length of hospital stay, presence of recurrence, pain in the first postoperative week, and time to complete epithelialization were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with pilonidal sinus disease in our hospital between November 2021 and November 2022

Exclusion Criteria:

* Patients under 18 years of age
* Acute pilonidal abcess
* Recurrent disease
* Anemic patients (Hg < 10 mg/dl)
* Thrombocytopenic patients (Plt˂10⁶/ml)
* Patients with a history of radiotherapy-chemotherapy
* Diabetes Mellitus
* Patients using steroids

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-01 (Actual)

PRIMARY OUTCOMES:
Platelet rich plasma accelerate the epithelialization of the wound after pilonidal sinus surgery | up to two months
  After the application of PRP the patients examined at the postoperative 2-4-6-10-15-20-25-30-35-40-45-50-55 days for the wound closure. The day of total epithelialization was noted.

SECONDARY OUTCOMES:
infection | up to two months
  presence of infection after surgery.
hematoma | up to two months
  presence of hematoma after surgery.
Pain intensity | up tp two months
  Pain intensity of patients measured by Visual analogue scale (VAS) score. 0 represents "no pain" and 10 "pain as bad as it could possibly be"
recurrence | up to two months
  Recurrence of the pilonidal disease of the patient is presence of pits in the previous surgical area and also presence a tender mass or sinus draining mucoid, purulent, and/or bloody fluid

CONTACTS AND LOCATIONS:
Locations (1):
- Diskapi Yildirim Beyazit Education And Research Hospital, Ankara, Altındag, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No